CLINICAL TRIAL: NCT01049451
Title: Comparison of Monthly Pulse ACTH (Acthar Gel) Therapy With Methylprednisolone (MP, Solumedrol) for Long-Term Treatment of Multiple Sclerosis (MS) as an Add on Therapy to Beta-interferons (Avonex, Betaseron or Rebif)
Brief Title: Pulse ACTH vs. MP for MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Regina Berkovich, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACTH-001; IND 104,973 (Registry Identifier: IND 104,973)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; ACTH; Steroids
MeSH Terms: conditions — Multiple Sclerosis | interventions — Adrenocorticotropic Hormone; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACTH IM monthly (Experimental): Subjects assigned to the ACTH arm will receive ACTH (Acthar gel) as intramuscular (IM) injections once a day for 3 consecutive days on a monthly basis, for 12 consecutive months. The dosage of ACTH will be 80 units per injection, for a total of 240 units over the three day period.
  Interventions: Drug: ACTH
- MP IV monthly (Active Comparator): Subjects assigned to the MP arm will receive intravenous (IV) infusions of 1 gram of MP once a month for 12 months.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: ACTH — Subjects assigned to the ACTH arm will receive ACTH (Acthar gel) as intramuscular (IM) injections once a day for 3 consecutive days on a monthly basis, for 12 consecutive months. The dosage of ACTH will be 80 units per injection, for a total of 240 units over the three day period.
  Other Names: Acthar Gel
  Arms: ACTH IM monthly
Drug: Methylprednisolone — Subjects assigned to the MP arm will receive intravenous (IV) infusions of 1 gram of MP once a month for 12 months
  Other Names: Solumedrol
  Arms: MP IV monthly

SUMMARY:
We hypothesize that corticotropin or adrenocorticotrophic hormone (ACTH), administered as Acthar Gel® (MANUFACTURER NAME) is effective in the control of clinical disease activity as a pulse therapy for relapsing-remitting MS when added to standard treatment with beta-interferon.

We wish to determine whether ACTH, when administered as clustered monthly intramuscular injections (monthly pulse therapy) as add-on to beta-interferons, may be a safe and effective alternative to monthly pulse therapy with MP. In addition, we hypothesize that pulse therapy with ACTH alters immune function to favor a regulatory, rather than a pro-inflammatory T cell environment.

DETAILED DESCRIPTION:
Please see the final manuscript

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite multiple sclerosis defined by McDonald Criteria.
2. Between 18-65 years of age.
3. Subject must able to understand and sign the IRB- approved informed consent form prior to the performance of any study-specific procedures and is willing to comply with the required scheduling and assessments of the protocol, including self-administration of study drug (if assigned to the ACTH arm).
4. Subjects who are women of childbearing potential, must have a negative serum pregnancy test at the screening visit, and must be willing to practice a reliable birth-control method.
5. Subjects must have at least one MS relapse within last year and/or at least one new T2 or Gadolinium-enhanced lesion on MRI while on stable interferon therapy.
6. EDSS (Expanded Disability Status Scale) score of 3.0 - 6.5
7. Currently on one of the approved beta-interferon drugs (Avonex, Betaseron, or Rebif) for a minimum of 6 months.

Exclusion Criteria:

1. Women who are either pregnant or breastfeeding, and women of child-bearing potential (defined as not surgically sterile or at least two years post menopausal) who are not using one of the following birth control methods: tubal ligation, implantable contraception device, oral, patch, injectable or transdermal contraceptive, barrier method or sexual activity restricted to vasectomized partner.
2. Uncontrolled hypertension, clinically significant cardiac arrhythmias, gastrointestinal ulcer, uncontrolled diabetes mellitus, osteoporosis, any stage of renal failure, psychiatric disorders or any other clinically significant general health conditions that may interfere with the trial participation.
3. Subject has a history of drug or alcohol abuse within the past year.
4. Subject had corticosteroid treatment within last 90 days.
5. Subject started new medication within last 30 days.
6. Subject is on Tysabri treatment presently or within 6 months of screening.
7. Subject is on Novantrone, Cellcept, Rituxan or other chemotherapeutic treatment presently or within 6 months of screening.
8. Subject is a participant in another research project.
9. Subject has contraindications for either ACTH or MP administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate | 15 months study: 12 months treatment and 3 months follow up

SECONDARY OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC), Expanded Disability Status Scale score (EDSS) and Multiple Sclerosis Quality of Life (MSQOL), peripheral blood lymphocytes measure for regulatory immune activities. | 15 months: 12 months treatmen and 3 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Regina R Berkovich, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC MS Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided